CLINICAL TRIAL: NCT03343626
Title: A Phase 1, Randomized, Observer-Blind, Placebo-Controlled, Safety, Immunogenicity, and Dose Ranging Study of Purified Inactivated Zika Virus Vaccine (PIZV) Candidate in Flavivirus Naïve and Primed Healthy Adults Aged 18 to 49 Years
Brief Title: Safety, Immunogenicity, and Dose Ranging Study of Inactivated Zika Virus Vaccine in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ZIK-101; U1111-1201-5778 (Registry Identifier: WHO)
Record Dates: First submitted 2017-11-13; First posted 2017-11-17 (Actual); Results first posted 2022-02-11 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2021-11

CONDITIONS: Virus, Zika; Zika Virus Disease; Flavivirus Infections; Healthy Participants
Keywords: Drug therapy
MeSH Terms: conditions — Zika Virus Infection; Flavivirus Infections

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Flavivirus-naïve Cohort: Placebo (Placebo Comparator): Placebo injection, intramuscular (IM), once on Day 1 (first dose) and Day 29 (second dose).
  Interventions: Drug: Placebo
- Flavivirus-naïve Cohort: PIZV 2 mcg (Low Dose) (Experimental): PIZV 0.5 mL, 2 mcg antigen, IM injection, once on Day 1 (first dose) and Day 29 (second dose).
  Interventions: Biological: PIZV
- Flavivirus-naïve Cohort: PIZV 5 mcg (Medium Dose) (Experimental): PIZV 0.5 mL, 5 mcg antigen, IM injection, once on Day 1 (first dose) and Day 29 (second dose).
  Interventions: Biological: PIZV
- Flavivirus-naïve Cohort: PIZV 10 mcg (High Dose) (Experimental): PIZV 0.5 mL, 10 mcg antigen, IM injection, once on Day 1 (first dose) and Day 29 (second dose).
  Interventions: Biological: PIZV
- Flavivirus-primed Cohort: Placebo (Placebo Comparator): Placebo injection, IM, once on Day 1 (first dose) and Day 29 (second dose).
  Interventions: Drug: Placebo
- Flavivirus-primed Cohort: PIZV 2 mcg (Low Dose) (Experimental): PIZV 0.5 mL, 2 mcg antigen, IM injection, once on Day 1 (first dose) and Day 29 (second dose).
  Interventions: Biological: PIZV
- Flavivirus-primed Cohort: PIZV 5 mcg (Medium Dose) (Experimental): PIZV 0.5 mL, 5 mcg antigen, IM injection, once on Day 1 (first dose) and Day 29 (second dose).
  Interventions: Biological: PIZV
- Flavivirus-primed Cohort: PIZV 10 mcg (High dose) (Experimental): PIZV 0.5 mL, 10 mcg antigen, IM injection, once on Day 1 (first dose) and Day 29 (second dose).
  Interventions: Biological: PIZV

INTERVENTIONS:
Drug: Placebo — Placebo (normal saline (0.9% NaCl) IM injection.
  Arms: Flavivirus-naïve Cohort: Placebo; Flavivirus-primed Cohort: Placebo
Biological: PIZV — Purified inactivated Zika virus vaccine with aluminum hydroxide adjuvant IM injection.
  Other Names: TAK-426
  Arms: Flavivirus-naïve Cohort: PIZV 10 mcg (High Dose); Flavivirus-naïve Cohort: PIZV 2 mcg (Low Dose); Flavivirus-naïve Cohort: PIZV 5 mcg (Medium Dose); Flavivirus-primed Cohort: PIZV 10 mcg (High dose); Flavivirus-primed Cohort: PIZV 2 mcg (Low Dose); Flavivirus-primed Cohort: PIZV 5 mcg (Medium Dose)

SUMMARY:
The purpose of this study is to describe the safety, tolerability and immunogenicity of two doses of purified inactivated Zika virus vaccine (PIZV) given 28 days apart. Three different vaccine doses containing different protein concentrations (2, 5 or 10 microgram [mcg]) each, will be given as 2 dose schedule to flavivirus naive and primed healthy adults. Participants will be followed for 7 days post each dose for tolerability and up to 6 months post dose 2 for safety. Immunogenicity assessment will be performed at 28 days post each dose and 6 months post dose 2. In addition, the selected dose group and control group will be followed till 24 months post dose 2 for safety and persistence of immunity.

DETAILED DESCRIPTION:
The vaccine being tested in this study is called PIZV or TAK-426 adjuvanted with aluminum hydroxide. The Zika virus vaccine is being tested to provide safety and immunogenicity data to enable the vaccine to be further developed clinically.

The study will enroll approximately 240 participants. Participants will be randomly assigned (by chance, like flipping a coin) to one of the four groups-which will remain undisclosed to the study observer:

* Placebo
* PIZV: 2 microgram (mcg) Low Dose
* PIZV: 5 mcg Medium Dose
* PIZV: 10 mcg High Dose

All participants will be administered either placebo or PIZV by intramuscular (IM) injection into the middle third of the deltoid muscle, preferably in the non-dominant arm on Days 1 (Visit 1) and 29 (Visit 4).

This multi-center trial will be conducted in the United States and Puerto Rico. The overall time to participate in this study is up to 25 months. Participants will make multiple visits to the clinic on Days 1, 8, 29, 36, 57, 211, 393 and will be contacted by telephone on Day 133 (Visit 7) and Day 575 (Visit 9) and also visit the clinic on Day 757 (Visit 11) depending on the study arm, for a final follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who are in good health at the time of entry into the trial as determined by medical history, physical examination (including vital signs) and eligibility screening tests (hematology, biochemistry and urinalysis) and clinical judgment of the investigator. Vital signs must be within normal limits (ie, below Grade 1 as specified in the Food and Drug Administration [FDA] Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers). Screening tests must be within normal limits or not be above Grade 1 as defined in the FDA Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers.
2. Participants who can comply with trial procedures and are available for the duration of follow-up.
3. All female participants must be willing to undergo serum beta human chorionic gonadotropin (B-hCG) pregnancy test and must test negative by urine pregnancy test prior to each study vaccination.

Exclusion Criteria:

1. Participants and participants' partners with confirmed Zika virus (ZIKV) infection by self-report.
2. Traveling to flavivirus endemic countries or flavivirus endemic regions of the United States (US) or US territories*, within 4 weeks prior to screening or planned travel through to Visit 6 (applicable only to participants to be enrolled into the flavivirus naïve cohort).

   a. Centers for Disease Control and Prevention (CDC) website define the information about the flavivirus endemic countries and US regions and territories.
3. Known hypersensitivity or allergy to any of the vaccine candidate components (including excipients of the investigational vaccine or placebo).
4. Has any history of progressive or severe neurologic disorder, seizure disorder or neuro-inflammatory disease (example, Guillain-Barré syndrome).
5. Known or suspected impairment/alteration of immune function, including:

   * Chronic use of oral steroids (equivalent to 20 milligram per day [mg/day] prednisone greater than or equal to [>=] 12 weeks / >= 2 milligram per kilogram [mg/kg] body weight / day prednisone >= 2 weeks) within 60 days prior to Day 1 (use of inhaled, intranasal, or topical corticosteroids is allowed).
   * Receipt of parenteral steroids (equivalent to 20 mg/day prednisone >= 12 weeks / >= 2 mg/kg body weight / day prednisone >= 2 weeks) within 60 days prior to Day 1.
   * Receipt of immunostimulants within 60 days prior to Day 1.
   * Receipt of parenteral, epidural or intra-articular immunoglobulin preparation, blood products, and/or plasma derived products within 3 months prior to Day 1 or planned during the full length of the trial. In addition, participants must be advised not to donate blood during the study period.
   * Known Human Immunodeficiency Virus (HIV) infection or HIV-related disease.
   * Genetic immunodeficiency.
6. Has known current or chronic hepatitis B and/or hepatitis C infections.
7. Has abnormalities of spleen or thymic function.
8. Has a known bleeding diathesis, or any condition that may be associated with a prolonged bleeding time.
9. Individuals participating in any clinical trial with another investigational product, including ZIKV vaccine clinical trial within 30 days prior to first trial visit or intent to participate in another clinical trial at any time during the conduct of this trial.
10. Individuals who received any other vaccines within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to enrollment in this trial or who are planning to receive any vaccine within 28 days of investigational vaccine/placebo administration.
11. Female participants who are pregnant or breastfeeding, or are planning to become pregnant.
12. Any positive or indeterminate pregnancy test.
13. If female participant of childbearing potential, sexually active, and who has not used any of the "acceptable contraceptive methods" for at least 2 months prior to trial entry:

    * "Of childbearing potential" is defined as status post onset of menarche and not meeting any of the following conditions: menopausal for at least 2 years without any other alternative medical cause (as confirmed by a healthcare professional), status after bilateral tubal ligation for at least 1 year, status after bilateral oophorectomy, or status after hysterectomy.
    * Acceptable birth control methods are defined as one or more of the following:

      * Hormonal contraceptive (such as oral, injection, transdermal patch, implant, cervical ring).
      * Barrier (condom with spermicide or diaphragm with spermicide) each and every time during intercourse.
      * Intrauterine device.
      * Monogamous relationship with vasectomized partner. Partner must have been vasectomized for at least six months prior to the participants' trial entry.
14. If female participant of childbearing potential and sexually active, refusal to use an "acceptable contraceptive method" from trial entry through 2 months after the last dose of investigational vaccine/placebo. In addition female participants of childbearing potential must be advised not to donate ova during this period.
15. To avoid sexual transmission of ZIKV from natural exposure: Refusal to use latex condoms correctly and consistently by sexually active participants even if other contraceptive measures are used from signing the informed consent form (ICF) through the end of the trial. Male participants must be advised not to donate sperm during this period.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 271 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2018-12-28 (Actual); Study Completion 2020-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (9):
- United States (7):
  - Clinical Research of South Florida, Coral Gables, Florida
  - Miami Research Associates, Miami, Florida
  - AppleMed Research, Miami, Florida
  - Johnson County Clin-Trials, Lenexa, Kansas
  - Regional Clinical Research Inc., Endwell, New York
  - Rochester Clinical Research, Rochester, New York
  - Tekton Research, Austin, Texas
- Puerto Rico (2):
  - Puerto Rico Clinical and Translational Research Consortium, San Juan, PR
  - Ponce Medical School Foundation, Santurce, PR

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Acosta CJ, Diaz C, Nordio F, Han HH, Moss KJ, Bohning K, Kumar P, Liu M, Patel H, Pacciarini F, Mwangi V, Walter E, Powell TD, El Sahly HM, Baldwin WR, Santangelo J, Anderson EJ, Dubin G. Persistence of Immunogenicity of a Purified Inactivated Zika Virus Vaccine Candidate in Healthy Adults: 2 Years of Follow-up Compared With Natural Infection. J Infect Dis. 2023 May 29;227(11):1303-1312. doi: 10.1093/infdis/jiac482. PMID 36484441
- [Derived] Han HH, Diaz C, Acosta CJ, Liu M, Borkowski A. Safety and immunogenicity of a purified inactivated Zika virus vaccine candidate in healthy adults: an observer-blind, randomised, phase 1 trial. Lancet Infect Dis. 2021 Sep;21(9):1282-1292. doi: 10.1016/S1473-3099(20)30733-7. Epub 2021 May 18. PMID 34019802

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants, aged >=18 to <=49 years, were enrolled in this Phase 1 study in 9 sites in the United States and Puerto Rico from 13 November 2017 to 24 November 2020.
Pre-assignment Details: Flavivirus (FV) status was determined using a Luminex assay targeting 13 FV. FV-naïve participants with median fluorescent intensity (MFI) below that assigned for negative cut-off were first enrolled in FV-naïve Cohort in ratio 1:1:1:1 to receive either placebo or purified inactivated Zika virus vaccine (PIZV). After positive recommendation from data monitoring committee, FV-primed participants, with MFI>500 were enrolled in FV-primed Cohort in ratio 1:1:1:1 to receive either placebo or PIZV.
Period: Overall Study
Arm/Group | Flavivirus-naïve Cohort: Placebo | Flavivirus-naïve Cohort: PIZV 2 mcg (Low Dose) | Flavivirus-naïve Cohort: PIZV 5 mcg (Medium Dose) | Flavivirus-naïve Cohort: PIZV 10 mcg (High Dose) | Flavivirus-primed Cohort: Placebo | Flavivirus-primed Cohort: PIZV 2 mcg (Low Dose) | Flavivirus-primed Cohort: PIZV 5 mcg (Medium Dose) | Flavivirus-primed Cohort: PIZV 10 mcg (High Dose)
Started | 31 | 31 | 31 | 32 | 36 | 37 | 37 | 36
Safety Analysis Set (Safety Analysis Set included all participants who received at least one (1) dose of PIZV or placebo.) | 31 | 31 | 31 | 32 | 36 | 37 | 37 | 36
Full Analysis Set (Full Analysis Set (FAS) included all randomized participants who had received at least one dose of the investigational vaccine/placebo and had provided valid Baseline and at least one post-vaccination serology result.) | 30 | 28 | 31 | 30 | 34 | 34 | 34 | 34
Per Protocol Set (Per-Protocol Set (PPS) included participants in the FAS who had no major protocol violations (relevant for the analysis, primary immunogenicity assessment or persistence assessment).) | 28 | 25 | 29 | 30 | 34 | 33 | 34 | 33
Completed | 25 | 26 | 29 | 24 | 29 | 32 | 32 | 25
Not Completed | 6 | 5 | 2 | 8 | 7 | 5 | 5 | 11
Not completed — Lost to Follow-up | 4 | 3 | 2 | 5 | 4 | 4 | 4 | 7
Not completed — Withdrawal of Consent | 2 | 1 | 0 | 3 | 3 | 1 | 1 | 2
Not completed — Reason not Specified | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Data Entry Error | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who received at least one (1) dose of PIZV or placebo.
Groups:
- Total: Total of all reporting groups
Arm/Group | Flavivirus-naïve Cohort: Placebo | Flavivirus-naïve Cohort: PIZV 2 mcg (Low Dose) | Flavivirus-naïve Cohort: PIZV 5 mcg (Medium Dose) | Flavivirus-naïve Cohort: PIZV 10 mcg (High Dose) | Flavivirus-primed Cohort: Placebo | Flavivirus-primed Cohort: PIZV 2 mcg (Low Dose) | Flavivirus-primed Cohort: PIZV 5 mcg (Medium Dose) | Flavivirus-primed Cohort: PIZV 10 mcg (High Dose) | Total
Number analyzed (Participants) | 31 | 31 | 31 | 32 | 36 | 37 | 37 | 36 | 271
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.7 (8.93) | 34.9 (9.52) | 35.8 (8.86) | 34.1 (8.50) | 34.7 (8.20) | 35.5 (8.71) | 37.0 (8.89) | 35.4 (8.45) | 35.5 (8.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 16 | 18 | 14 | 21 | 18 | 26 | 24 | 158
  Male | 10 | 15 | 13 | 18 | 15 | 19 | 11 | 12 | 113
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2 | 4 | 36 | 36 | 36 | 35 | 151
  Not Hispanic or Latino | 30 | 30 | 29 | 28 | 0 | 1 | 0 | 1 | 119
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
  Black or African American | 6 | 5 | 3 | 4 | 6 | 4 | 7 | 10 | 45
  White | 23 | 26 | 26 | 27 | 27 | 31 | 30 | 25 | 215
  More than one race | 0 | 0 | 2 | 1 | 1 | 1 | 0 | 1 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States of America | 31 | 31 | 31 | 32 | 21 | 21 | 21 | 21 | 209
  Puerto Rico | 0 | 0 | 0 | 0 | 15 | 16 | 16 | 15 | 62
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI is calculated as weight (kg) divided by square of height (m^2).
  kg/m^2 | 27.921 (4.2049) | 27.527 (4.7632) | 27.541 (3.7165) | 26.750 (3.6511) | 27.398 (3.5244) | 27.054 (4.7105) | 26.982 (4.1240) | 28.072 (4.4735) | 27.398 (4.1433)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Solicited Local Injection Site Reactions by Severity Within 7 Days After Dose 1 of PIZV or Placebo
Description: Solicited local AEs (at injection site) were collected by participants using diary cards within 7 days after first vaccination and included pain (none, mild: no interference with daily activity, moderate: interference with daily activity with or without treatment and severe: prevents daily activity with or without treatment), erythema (<25 mm, mild: >=25 to- <=50 mm, moderate: >50 to <=100 mm, severe: >100 mm), and swelling and induration (<25 mm, mild: >=25 to <=-50 mm, moderate: >50 to <=100 mm, severe: >100 mm). Only categories for which there was at least 1 participant are reported.
Time Frame: Within 7 days after Dose 1 (Day 8)
Population: Safety Analysis Set included all randomized participants who received at least one (1) dose of PIZV or placebo. Overall number of participants are the number of participants with data available for analyses.
Measure: Number; unit: percentage of participants
Arm/Group | Flavivirus-naïve Cohort: Placebo | Flavivirus-naïve Cohort: PIZV 2 mcg (Low Dose) | Flavivirus-naïve Cohort: PIZV 5 mcg (Medium Dose) | Flavivirus-naïve Cohort: PIZV 10 mcg (High Dose) | Flavivirus-primed Cohort: Placebo | Flavivirus-primed Cohort: PIZV 2 mcg (Low Dose) | Flavivirus-primed Cohort: PIZV 5 mcg (Medium Dose) | Flavivirus-primed Cohort: PIZV 10 mcg (High Dose)
Number analyzed (Participants) | 30 | 30 | 31 | 31 | 36 | 33 | 36 | 35
percentage of participants
  Pain, Mild | 13.3 | 30.0 | 32.3 | 38.7 | 8.3 | 33.3 | 30.6 | 34.3
  Pain, Moderate | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 9.1 | 8.3 | 2.9
  Pain, Severe | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 3.0 | 0.0 | 0.0
  Erythema, <25 mm | 0.0 | 0.0 | 0.0 | 3.2 | 5.6 | 3.0 | 2.8 | 0.0
  Induration, <25 mm | 0.0 | 0.0 | 9.7 | 6.5 | 0.0 | 3.0 | 5.6 | 0.0
  Swelling, <25 mm | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 6.1 | 5.6 | 2.9

2. Primary Outcome: Percentage of Participants With Solicited Local Injection Site Reactions by Severity Within 7 Days After Dose 2 of PIZV or Placebo
Description: Solicited local AEs (at injection site) were collected by participants using diary cards within 7 days after first vaccination and included pain (none, mild: no interference with daily activity, moderate: interference with daily activity with or without treatment and severe: prevents daily activity with or without treatment), erythema (<25 mm, mild: >=25 to <=50 mm, moderate: >50 to <=100 mm, severe: >100 mm), and swelling and induration (<25 mm, mild: >=25 to <=50 mm, moderate: >50 to <=100 mm, severe: >100 mm). Only categories for which there was at least 1 participant are reported.
Time Frame: Within 7 days after Dose 2 (Day 36)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Flavivirus-naïve Cohort: Placebo | Flavivirus-naïve Cohort: PIZV 2 mcg (Low Dose) | Flavivirus-naïve Cohort: PIZV 5 mcg (Medium Dose) | Flavivirus-naïve Cohort: PIZV 10 mcg (High Dose) | Flavivirus-primed Cohort: Placebo | Flavivirus-primed Cohort: PIZV 2 mcg (Low Dose) | Flavivirus-primed Cohort: PIZV 5 mcg (Medium Dose) | Flavivirus-primed Cohort: PIZV 10 mcg (High Dose)
Number analyzed (Participants) | 28 | 27 | 30 | 30 | 33 | 32 | 32 | 34
percentage of participants
  Pain, Mild | 14.3 | 29.6 | 30.0 | 36.7 | 18.2 | 21.9 | 21.9 | 20.6
  Pain, Moderate | 0.0 | 0.0 | 6.7 | 3.3 | 0.0 | 0.0 | 6.3 | 8.8
  Erythema, <25 mm | 3.6 | 0.0 | 3.3 | 3.3 | 0.0 | 3.1 | 3.1 | 2.9
  Erythema, Mild | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 3.2 | 0.0 | 0.0
  Induration, <25 mm | 0.0 | 0.0 | 3.3 | 0.0 | 0.0 | 0.0 | 3.1 | 2.9
  Swelling, <25 mm | 0.0 | 0.0 | 6.7 | 0.0 | 0.0 | 0.0 | 0.0 | 5.9
  Swelling, Mild | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 3.1 | 0.0 | 0.0

3. Primary Outcome: Percentage of Participants With Solicited Systemic Adverse Events (AEs) by Severity Within 7 Days After Dose 1 of PIZV or Placebo
Description: Solicited systemic AEs included fever, headache, fatigue, malaise, arthralgia, and myalgia that occurred within 7 days of first vaccination. Solicited systemic AEs (headache, fatigue, malaise, arthralgia, and myalgia) was graded from 0 to 3 by severity; where 0=None, 1=Mild: No interference with daily activity, 2=Moderate: Interference with daily activity, 3=Severe: Prevents daily activity; A systemic AE of fever (defined as ≥38°C or ≥100.4°F) was graded from 1 to 4 by severity; where 1=Mild: 38.0-38.4°C, 2=Moderate: 38.5-38.9°C, 3=Severe: 39.0-40°C, and 4=Potentially life threatening:>40°C. Only categories for which there was at least 1 participant are reported.
Time Frame: Within 7 days after Dose 1 (Day 8)
Population: Safety Analysis Set included all randomized participants who received at least one (1) dose of PIZV or placebo. Number analyzed is the number of participants with data available for analyses in the specific category.
Measure: Number; unit: percentage of participants
Arm/Group | Flavivirus-naïve Cohort: Placebo | Flavivirus-naïve Cohort: PIZV 2 mcg (Low Dose) | Flavivirus-naïve Cohort: PIZV 5 mcg (Medium Dose) | Flavivirus-naïve Cohort: PIZV 10 mcg (High Dose) | Flavivirus-primed Cohort: Placebo | Flavivirus-primed Cohort: PIZV 2 mcg (Low Dose) | Flavivirus-primed Cohort: PIZV 5 mcg (Medium Dose) | Flavivirus-primed Cohort: PIZV 10 mcg (High Dose)
Number analyzed (Participants) | 31 | 31 | 31 | 32 | 36 | 37 | 37 | 36
percentage of participants
  Fever, Mild: number analyzed (Participants) | 31 | 31 | 31 | 32 | 35 | 32 | 37 | 36
  Fever, Mild | 3.3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 2.8 | 0.0
  Fever, Moderate: number analyzed (Participants) | 31 | 31 | 31 | 32 | 35 | 32 | 37 | 36
  Fever, Moderate | 0.0 | 0.0 | 0.0 | 3.2 | 0.0 | 0.0 | 0.0 | 0.0
  Headache, Mild | 20.0 | 13.3 | 19.4 | 12.9 | 11.1 | 12.1 | 13.9 | 11.4
  Headache, Moderate | 13.3 | 3.3 | 6.5 | 0.0 | 2.8 | 3.0 | 5.6 | 2.9
  Headache, Severe | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 2.8 | 2.9
  Fatigue, Mild | 16.7 | 16.7 | 16.1 | 25.8 | 16.7 | 6.1 | 25.0 | 17.1
  Fatigue, Moderate | 6.7 | 6.7 | 3.2 | 6.5 | 8.3 | 3.0 | 0.0 | 0.0
  Arthralgia, Mild | 3.3 | 0.0 | 3.2 | 6.5 | 8.3 | 12.1 | 11.1 | 5.7
  Arthralgia, Moderate | 0.0 | 3.3 | 0.0 | 3.2 | 0.0 | 0.0 | 0.0 | 0.0
  Myalgia, Mild | 6.7 | 6.7 | 16.1 | 12.9 | 19.4 | 12.1 | 13.9 | 8.6
  Myalgia, Moderate | 3.3 | 3.3 | 0.0 | 0.0 | 0.0 | 2.7 | 0.0 | 0.0
  Myalgia, Severe | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 3.0 | 0.0 | 2.9
  Malaise, Mild | 6.7 | 3.3 | 3.2 | 12.9 | 19.4 | 12.1 | 16.7 | 22.9
  Malaise, Moderate | 6.7 | 3.3 | 3.2 | 0.0 | 2.8 | 0.0 | 0.0 | 0.0

4. Primary Outcome: Percentage of Participants With Solicited Systemic AEs by Severity Within 7 Days After Dose 2 of PIZV or Placebo
Description: as for outcome 3
Time Frame: Within 7 days after Dose 2 (Day 36)
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Flavivirus-naïve Cohort: Placebo | Flavivirus-naïve Cohort: PIZV 2 mcg (Low Dose) | Flavivirus-naïve Cohort: PIZV 5 mcg (Medium Dose) | Flavivirus-naïve Cohort: PIZV 10 mcg (High Dose) | Flavivirus-primed Cohort: Placebo | Flavivirus-primed Cohort: PIZV 2 mcg (Low Dose) | Flavivirus-primed Cohort: PIZV 5 mcg (Medium Dose) | Flavivirus-primed Cohort: PIZV 10 mcg (High Dose)
Number analyzed (Participants) | 31 | 31 | 31 | 32 | 36 | 37 | 37 | 36
percentage of participants
  Fever, Mild: number analyzed (Participants) | 28 | 31 | 31 | 32 | 36 | 31 | 31 | 36
  Fever, Mild | 3.2 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Fever, Severe: number analyzed (Participants) | 28 | 31 | 31 | 32 | 36 | 31 | 31 | 36
  Fever, Severe | 3.2 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 6.4 | 0.0
  Headache, Mild | 6.9 | 14.8 | 0.0 | 16.7 | 6.1 | 6.3 | 12.5 | 2.9
  Headache, Moderate | 3.4 | 0.0 | 3.3 | 3.3 | 3.3 | 0.0 | 0.0 | 8.8
  Headache, Severe | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 3.1 | 0.0
  Fatigue, Mild | 13.8 | 11.1 | 3.3 | 13.3 | 9.1 | 3.1 | 9.4 | 11.8
  Fatigue, Moderate | 6.9 | 0.0 | 3.3 | 3.3 | 0.0 | 0.0 | 3.1 | 2.9
  Arthralgia, Mild | 0.0 | 7.4 | 0.0 | 0.0 | 0.0 | 9.4 | 3.1 | 2.9
  Arthralgia, Moderate | 3.4 | 0.0 | 0.0 | 3.3 | 0.0 | 0.0 | 3.1 | 2.9
  Arthralgia, Severe | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 3.1 | 0.0
  Myalgia, Mild | 0.0 | 7.4 | 3.3 | 3.3 | 9.1 | 12.5 | 6.3 | 2.9
  Myalgia, Moderate | 6.9 | 0.0 | 0.0 | 3.3 | 0.0 | 0.0 | 0.0 | 5.9
  Myalgia, Severe | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 3.1 | 2.9
  Malaise, Mild | 3.4 | 0.0 | 0.0 | 6.7 | 12.1 | 3.1 | 6.3 | 2.9
  Malaise, Moderate | 3.4 | 0.0 | 0.0 | 3.3 | 3.0 | 0.0 | 3.1 | 5.9
  Malaise, Severe | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 3.1 | 0.0

5. Primary Outcome: Percentage of Participants Who Experienced at Least One Non-serious Unsolicited AE Within 28 Days After Dose 1 of PIZV or Placebo
Description: An AE was defined as any untoward medical occurrence in participants administered a trial vaccine; it does not necessarily have to have a causal relationship with trial vaccine administration.
Time Frame: Within 28 days after Dose 1 (Day 29)
Population: Safety Analysis Set included all randomized participants who received at least one (1) dose of PIZV or placebo.
Measure: Number; unit: percentage of participants
Arm/Group | Flavivirus-naïve Cohort: Placebo | Flavivirus-naïve Cohort: PIZV 2 mcg (Low Dose) | Flavivirus-naïve Cohort: PIZV 5 mcg (Medium Dose) | Flavivirus-naïve Cohort: PIZV 10 mcg (High Dose) | Flavivirus-primed Cohort: Placebo | Flavivirus-primed Cohort: PIZV 2 mcg (Low Dose) | Flavivirus-primed Cohort: PIZV 5 mcg (Medium Dose) | Flavivirus-primed Cohort: PIZV 10 mcg (High Dose)
Number analyzed (Participants) | 31 | 31 | 31 | 32 | 36 | 37 | 37 | 36
percentage of participants | 29.0 | 19.4 | 29.0 | 9.4 | 22.2 | 21.6 | 21.6 | 16.7

6. Primary Outcome: Percentage of Participants Who Experienced at Least One Non-serious Unsolicited AE Within 28 Days After Dose 2 of PIZV or Placebo
Description: An AE was defined as any untoward medical occurrence in a clinical investigation participants administered a trial vaccine; it does not necessarily have to have a causal relationship with trial vaccine administration.
Time Frame: Within 28 days after Dose 2 (Day 57)
Population: Safety Analysis Set included all randomized participants who received at least one (1) dose of PIZV or placebo.
Measure: Number; unit: percentage of participants
Arm/Group | Flavivirus-naïve Cohort: Placebo | Flavivirus-naïve Cohort: PIZV 2 mcg (Low Dose) | Flavivirus-naïve Cohort: PIZV 5 mcg (Medium Dose) | Flavivirus-naïve Cohort: PIZV 10 mcg (High Dose) | Flavivirus-primed Cohort: Placebo | Flavivirus-primed Cohort: PIZV 2 mcg (Low Dose) | Flavivirus-primed Cohort: PIZV 5 mcg (Medium Dose) | Flavivirus-primed Cohort: PIZV 10 mcg (High Dose)
Number analyzed (Participants) | 31 | 31 | 31 | 32 | 36 | 37 | 37 | 36
percentage of participants | 16.1 | 16.1 | 9.7 | 12.5 | 8.3 | 13.5 | 13.5 | 13.9

7. Primary Outcome: Percentage of Participants Who Experienced at Least One Serious Adverse Event (SAE) Within 28 Days After Dose 1 of PIZV or Placebo
Description: A SAE was defined as any untoward medical occurrence that: 1) results in death, 2) is life-threatening, 3) requires inpatient hospitalization or prolongation of existing hospitalization, 4) results in persistent or significant disability/incapacity, 5) leads to a congenital anomaly/birth defect in the offspring of the participant or 6) is an medically important event that satisfies any of the following: a) May require intervention to prevent items 1 through 5 above. b) May expose the participant to danger, even though the event is not immediately life threatening or fatal or does not result in hospitalization.
Time Frame: Within 28 days after Dose 1 (Day 29)
Population: Safety Analysis Set included all randomized participants who received at least one (1) dose of PIZV or placebo.
Measure: Number; unit: percentage of participants
Arm/Group | Flavivirus-naïve Cohort: Placebo | Flavivirus-naïve Cohort: PIZV 2 mcg (Low Dose) | Flavivirus-naïve Cohort: PIZV 5 mcg (Medium Dose) | Flavivirus-naïve Cohort: PIZV 10 mcg (High Dose) | Flavivirus-primed Cohort: Placebo | Flavivirus-primed Cohort: PIZV 2 mcg (Low Dose) | Flavivirus-primed Cohort: PIZV 5 mcg (Medium Dose) | Flavivirus-primed Cohort: PIZV 10 mcg (High Dose)
Number analyzed (Participants) | 31 | 31 | 31 | 32 | 36 | 37 | 37 | 36
percentage of participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 2.7 | 0.0 | 0.0

8. Primary Outcome: Percentage of Participants Who Experienced at Least One SAE Within 28 Days After Dose 2 of PIZV or Placebo
Description: as for outcome 7
Time Frame: Within 28 days after Dose 2 (Day 57)
Population: Safety Analysis Set included all randomized participants who received at least one (1) dose of PIZV or placebo.
Measure: Number; unit: percentage of participants
Arm/Group | Flavivirus-naïve Cohort: Placebo | Flavivirus-naïve Cohort: PIZV 2 mcg (Low Dose) | Flavivirus-naïve Cohort: PIZV 5 mcg (Medium Dose) | Flavivirus-naïve Cohort: PIZV 10 mcg (High Dose) | Flavivirus-primed Cohort: Placebo | Flavivirus-primed Cohort: PIZV 2 mcg (Low Dose) | Flavivirus-primed Cohort: PIZV 5 mcg (Medium Dose) | Flavivirus-primed Cohort: PIZV 10 mcg (High Dose)
Number analyzed (Participants) | 31 | 31 | 31 | 32 | 36 | 37 | 37 | 36
percentage of participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

9. Primary Outcome: Geometric Mean Titers (GMTs) of Neutralizing Antibody for Zika Virus (ZIKV) 28 Days After Dose 2 of PIZV or Placebo
Description: GMTs of neutralizing antibodies for ZIKV were measured by the Zika plaque reduction neutralization test (PRNT) test, by assessing the quantity of neutralizing antibodies that bind ZIKV in the assay. The assay results were reported as titers (reciprocal value of the dilution of the serum from the vaccinated individual that inhibits for 50% the plaque formation).
Time Frame: 28 days after Dose 2 (Day 57)
Population: Per-Protocol Set (PPS) included participants in the Full Analysis Set (FAS) who have no major protocol violations (relevant for the analysis, primary immunogenicity assessment or persistence assessment). Overall number of participants analyzed are the number of participants with data available for analyses.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Flavivirus-naïve Cohort: Placebo | Flavivirus-naïve Cohort: PIZV 2 mcg (Low Dose) | Flavivirus-naïve Cohort: PIZV 5 mcg (Medium Dose) | Flavivirus-naïve Cohort: PIZV 10 mcg (High Dose) | Flavivirus-primed Cohort: Placebo | Flavivirus-primed Cohort: PIZV 2 mcg (Low Dose) | Flavivirus-primed Cohort: PIZV 5 mcg (Medium Dose) | Flavivirus-primed Cohort: PIZV 10 mcg (High Dose)
Number analyzed (Participants) | 27 | 23 | 28 | 28 | 31 | 30 | 31 | 30
titer | 5.00 [NA to NA] — The upper and lower limit of 95% confidence interval were not available as the titers were below the limits of quantification. As prespecified in the study, the antibody titers below the specific Limit of detection (LOD)=10 was assigned median titer value equal to half of the LOD titer. | 1129.69 [749.38 to 1703.1] | 1992.33 [1401.28 to 2832.70] | 3689.89 [2676.75 to 5086.49] | 198.82 [91.73 to 430.97] | 597.63 [340.48 to 1049.00] | 1276.92 [806.00 to 2022.97] | 2590.54 [1649.18 to 4069.22]

10. Secondary Outcome: Percentage of Participants Who Experienced at Least One SAE During the Study
Description: as for outcome 7
Time Frame: From day of first vaccination (Day 1) up to end of the study (Day 757)
Population: Safety Analysis Set included all randomized participants who received at least one (1) dose of PIZV or placebo.
Measure: Number; unit: percentage of participants
Arm/Group | Flavivirus-naïve Cohort: Placebo | Flavivirus-naïve Cohort: PIZV 2 mcg (Low Dose) | Flavivirus-naïve Cohort: PIZV 5 mcg (Medium Dose) | Flavivirus-naïve Cohort: PIZV 10 mcg (High Dose) | Flavivirus-primed Cohort: Placebo | Flavivirus-primed Cohort: PIZV 2 mcg (Low Dose) | Flavivirus-primed Cohort: PIZV 5 mcg (Medium Dose) | Flavivirus-primed Cohort: PIZV 10 mcg (High Dose)
Number analyzed (Participants) | 31 | 31 | 31 | 32 | 36 | 37 | 37 | 36
percentage of participants | 3.2 | 3.2 | 0.0 | 6.3 | 2.8 | 5.4 | 0.0 | 11.1

11. Secondary Outcome: GMTs of Neutralizing Antibody for ZIKV 28 Days After Dose 1 and 6 Months After Dose 2
Description: GMTs of neutralizing antibodies for ZIKV were measured by Zika PRNT test, by assessing the quantity of neutralizing antibodies that bind ZIKV in the assay. The assay results were reported as titers (reciprocal value of the dilution of the serum from the vaccinated individual that inhibits for 50% the plaque formation).
Time Frame: 28 days after Dose 1 (Day 29); 6 months after Dose 2 (Day 211)
Population: PPS included participants in the FAS who have no major protocol violations (relevant for the analysis, primary immunogenicity assessment or persistence assessment). Number analyzed is the number of participants with data available for analysis at the given tlmepoint.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Flavivirus-naïve Cohort: Placebo | Flavivirus-naïve Cohort: PIZV 2 mcg (Low Dose) | Flavivirus-naïve Cohort: PIZV 5 mcg (Medium Dose) | Flavivirus-naïve Cohort: PIZV 10 mcg (High Dose) | Flavivirus-primed Cohort: Placebo | Flavivirus-primed Cohort: PIZV 2 mcg (Low Dose) | Flavivirus-primed Cohort: PIZV 5 mcg (Medium Dose) | Flavivirus-primed Cohort: PIZV 10 mcg (High Dose)
Number analyzed (Participants) | 28 | 25 | 29 | 30 | 34 | 33 | 34 | 33
titer
  Day 29 | 5.00 [NA to NA] — The upper and lower limit of 95% confidence interval were not available as the titers were below the limits of quantification. As prespecified in the study, the antibody titers below the specific Limit of detection (LOD)=10 was assigned median titer value equal to half of the LOD titer. | 41.28 [18.74 to 90.95] | 93.76 [44.34 to 198.30] | 291.41 [161.74 to 525.06] | 164.06 [77.37 to 347.88] | 513.62 [259.90 to 1015.03] | 1002.69 [566.72 to 1774.06] | 1572.58 [864.63 to 2860.20]
  Day 211: number analyzed (Participants) | 21 | 20 | 25 | 23 | 30 | 25 | 26 | 26
  Day 211 | 5.00 [NA to NA] — The upper and lower limit of 95% confidence interval were not available as the titers were below the limits of quantification. As prespecified in the study, the antibody titers below the specific Limit of detection (LOD)=10 was assigned median titer value equal to half of the LOD titer. | 151.24 [87.27 to 262.10] | 364.10 [237.97 to 557.08] | 613.28 [382.29 to 983.83] | 125.80 [48.02 to 329.55] | 258.44 [93.32 to 715.73] | 506.97 [228.56 to 1124.50] | 866.26 [445.59 to 1684.08]

12. Secondary Outcome: GMTs of Neutralizing Antibody for ZIKV 12 Months and 24 Months After Dose 2 in Applicable Groups
Description: GMTs of neutralizing antibodies for ZIKV were measured by Zika PRNT test, by assessing the quantity of neutralizing antibodies that bind ZIKV in the assay. The assay results were reported as titers (reciprocal value of the dilution of the serum from the vaccinated individual that inhibits for 50% the plaque formation). As prespecified in the protocol, only data for applicable groups (Placebo and PIZV 10 mcg who were followed beyond Day 211) were analyzed and reported at Days 393 and 757 for Flavivirus-naïve Cohort and Flavivirus-primed Cohort.
Time Frame: 12 months after Dose 2 (Day 393); 24 months after Dose 2 (Day 757)
Population: PPS included participants in the FAS who had no major protocol violations (relevant for the analysis, primary immunogenicity assessment or persistence assessment). Overall number of participants analyzed are the number of participants with data available for analyses. Number analyzed is the number of participants with data available for analysis at the given timepoint.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Flavivirus-naïve Cohort: Placebo | Flavivirus-naïve Cohort: PIZV 10 mcg (High Dose) | Flavivirus-primed Cohort: Placebo | Flavivirus-primed Cohort: PIZV 10 mcg (High Dose)
Number analyzed (Participants) | 28 | 30 | 34 | 31
titer
  Day 393: number analyzed (Participants) | 28 | 30 | 34 | 25
  Day 393 | 5.00 [NA to NA] — The upper and lower limit of 95% confidence interval were not available as the titers were below the limits of quantification. As prespecified in the study, the antibody titers below the specific Limit of detection (LOD)=10 was assigned median titer value equal to half of the LOD titer. | 413.71 [215.67 to 793.58] | 103.88 [39.85 to 270.78] | 505.10 [287.58 to 887.15]
  Day 757: number analyzed (Participants) | 19 | 16 | 27 | 21
  Day 757 | 18.48 [6.00 to 56.91] | 427.41 [171.06 to 1067.93] | 324.26 [131.54 to 799.36] | 149.68 [56.68 to 395.24]

13. Secondary Outcome: Percentage of Participants Seropositive for Neutralizing Antibodies Against PIZV 28 Days After Dose 1, 28 Days After Dose 2, and 6 Months After Dose 2
Description: Seropositive participants were defined as participants with detectable serum antibodies (tested positive at or above limit of detection, LOD) as measured by the neutralization assay.
Time Frame: 28 days after Dose 1 (Day 29); 28 days after Dose 2 (Day 57); 6 months after Dose 2 (Day 211)
Population: PPS included participants in the FAS who had no major protocol violations (relevant for the analysis, primary immunogenicity assessment or persistence assessment). Number analyzed is the number of participants with data available for analysis at the given timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Flavivirus-naïve Cohort: Placebo | Flavivirus-naïve Cohort: PIZV 2 mcg (Low Dose) | Flavivirus-naïve Cohort: PIZV 5 mcg (Medium Dose) | Flavivirus-naïve Cohort: PIZV 10 mcg (High Dose) | Flavivirus-primed Cohort: Placebo | Flavivirus-primed Cohort: PIZV 2 mcg (Low Dose) | Flavivirus-primed Cohort: PIZV 5 mcg (Medium Dose) | Flavivirus-primed Cohort: PIZV 10 mcg (High Dose)
Number analyzed (Participants) | 28 | 25 | 29 | 30 | 34 | 33 | 34 | 33
percentage of participants
  Day 29: number analyzed (Participants) | 28 | 25 | 28 | 28 | 34 | 31 | 34 | 33
  Day 29 | 0.0 [NA to NA] — Data for lower and upper limit of 95% CI was not estimable for this timepoint as the concentration were below the level of detection. | 72.00 [50.61 to 87.93] | 82.14 [63.11 to 93.94] | 96.43 [81.65 to 99.91] | 85.29 [68.94 to 95.05] | 96.77 [83.30 to 99.92] | 100.00 [89.72 to 100.00] | 100.00 [89.42 to 100.0]
  Day 57: number analyzed (Participants) | 27 | 23 | 28 | 28 | 31 | 30 | 31 | 30
  Day 57 | 0.0 [NA to NA] — Data for lower and upper limit of 95% CI was not estimable for this timepoint as the concentration were below the level of detection. | 100.00 [85.18 to 100.00] | 100.00 [87.66 to 100.00] | 100.00 [87.66 to 100.00] | 87.10 [70.17 to 96.37] | 96.67 [82.78 to 99.92] | 100.00 [88.78 to 100.00] | 100.00 [88.43 to 100.00]
  Day 211: number analyzed (Participants) | 21 | 20 | 25 | 23 | 30 | 25 | 26 | 26
  Day 211 | 0.0 [NA to NA] — Data for lower and upper limit of 95% CI was not estimable for this timepoint as the concentration were below the level of detection. | 100.00 [83.16 to 100.00] | 100.00 [86.28 to 100.0] | 100.00 [85.18 to 100.00] | 76.67 [57.72 to 90.07] | 84.00 [63.92 to 95.46] | 100.00 [86.77 to 100.00] | 100.00 [86.77 to 100.00]

14. Secondary Outcome: Percentage of Participants Seropositive for PIZV 12 Months and 24 Months After Dose 2 in Applicable Groups
Description: Seropositive participants were defined as participants with detectable serum antibodies (tested positive at or above limit of detection, LOD) as measured by the neutralization assay. As prespecified in the protocol, only data for applicable groups (Placebo and PIZV 10 mcg who were followed beyond Day 211) were analyzed and reported at Days 393 and 757 for Flavivirus-naïve Cohort and Flavivirus-primed Cohort.
Time Frame: 12 months after Dose 2 (Day 393); 24 months after Dose 2 (Day 757)
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Flavivirus-naïve Cohort: Placebo | Flavivirus-naïve Cohort: PIZV 10 mcg (High Dose) | Flavivirus-primed Cohort: Placebo | Flavivirus-primed Cohort: PIZV 10 mcg (High Dose)
Number analyzed (Participants) | 28 | 30 | 34 | 31
percentage of participants
  Day 393: number analyzed (Participants) | 23 | 21 | 32 | 25
  Day 393 | 0.00 [0.00 to 14.82] | 100.0 [83.89 to 100.0] | 65.63 [46.81 to 81.43] | 100.0 [86.28 to 100.0]
  Day 757: number analyzed (Participants) | 19 | 16 | 27 | 21
  Day 757 | 26.32 [9.15 to 51.20] | 93.75 [69.77 to 99.84] | 85.19 [66.27 to 95.81] | 76.19 [52.83 to 91.78]

15. Secondary Outcome: Percentage of Participants Seroconverted for PIZV 28 Days Post Dose 1 and 28 Days Post Dose 2
Description: Seroconverted participants were defined as participants at Baseline with detectable post-vaccination serum antibodies (test results are at or above LOD) and seropositive participants at Baseline with a four-fold increase in post-vaccination antibodies from Baseline, as measured by the neutralization assay.
Time Frame: 28 days after Dose 1 (Day 29); 28 days after Dose 2 (Day 57)
Population: Per-Protocol Set (PPS) included participants in the Full Analysis Set (FAS) who have no major protocol violations (relevant for the analysis, primary immunogenicity assessment or persistence assessment). Number analyzed is the number of participants with data available for analysis at the given tlmepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Flavivirus-naïve Cohort: Placebo | Flavivirus-naïve Cohort: PIZV 2 mcg (Low Dose) | Flavivirus-naïve Cohort: PIZV 5 mcg (Medium Dose) | Flavivirus-naïve Cohort: PIZV 10 mcg (High Dose) | Flavivirus-primed Cohort: Placebo | Flavivirus-primed Cohort: PIZV 2 mcg (Low Dose) | Flavivirus-primed Cohort: PIZV 5 mcg (Medium Dose) | Flavivirus-primed Cohort: PIZV 10 mcg (High Dose)
Number analyzed (Participants) | 28 | 25 | 29 | 30 | 34 | 33 | 34 | 33
percentage of participants
  Day 29: number analyzed (Participants) | 28 | 25 | 28 | 28 | 34 | 31 | 34 | 33
  Day 29 | 0.0 [NA to NA] — Data for lower and upper limit of 95% CI was not estimable for this timepoint as the concentration were below the level of detection. | 72.00 [50.61 to 87.93] | 82.14 [63.11 to 93.94] | 96.43 [81.65 to 99.91] | 2.94 [0.07 to 15.33] | 38.71 [21.85 to 57.81] | 50.00 [32.43 to 67.57] | 69.70 [51.29 to 84.41]
  Day 57: number analyzed (Participants) | 27 | 23 | 28 | 28 | 31 | 30 | 31 | 30
  Day 57 | 0.0 [NA to NA] — Data for lower and upper limit of 95% CI was not estimable for this timepoint as the concentration were below the level of detection. | 100.00 [85.18 to 100.0] | 100.00 [87.66 to 100.00] | 100.00 [87.66 to 100.0] | 6.45 [0.79 to 21.42] | 46.67 [28.34 to 65.67] | 54.84 [36.03 to 72.68] | 76.67 [57.72 to 90.07]

ADVERSE EVENTS:
Time Frame: All Cause Mortality and Serious Adverse Events: From day of first vaccination (Day 1) up to end of the study (Day 757); Non Serious Adverse Events: Up to 28 days (day of vaccination + 27 days) after administration of each vaccine dose on Day 1 and Day 29
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Flavivirus-naïve Cohort: Placebo | Flavivirus-naïve Cohort: PIZV 2 mcg (Low Dose) | Flavivirus-naïve Cohort: PIZV 5 mcg (Medium Dose) | Flavivirus-naïve Cohort: PIZV 10 mcg (High Dose) | Flavivirus-primed Cohort: Placebo | Flavivirus-primed Cohort: PIZV 2 mcg (Low Dose) | Flavivirus-primed Cohort: PIZV 5 mcg (Medium Dose) | Flavivirus-primed Cohort: PIZV 10 mcg (High Dose)
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/31 | 0/31 | 0/32 | 0/36 | 0/37 | 0/37 | 0/36
Serious Adverse Events (participants affected / at risk) | 1/31 | 1/31 | 0/31 | 2/32 | 1/36 | 2/37 | 0/37 | 4/36
Other Adverse Events (participants affected / at risk) | 4/31 | 3/31 | 3/31 | 4/32 | 5/36 | 5/37 | 7/37 | 8/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Flavivirus-naïve Cohort: Placebo (N=31) | Flavivirus-naïve Cohort: PIZV 2 mcg (Low Dose) (N=31) | Flavivirus-naïve Cohort: PIZV 5 mcg (Medium Dose) (N=31) | Flavivirus-naïve Cohort: PIZV 10 mcg (High Dose) (N=32) | Flavivirus-primed Cohort: Placebo (N=36) | Flavivirus-primed Cohort: PIZV 2 mcg (Low Dose) (N=37) | Flavivirus-primed Cohort: PIZV 5 mcg (Medium Dose) (N=37) | Flavivirus-primed Cohort: PIZV 10 mcg (High Dose) (N=36)
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Major depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adenomyosis (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Premature delivery (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Flavivirus-naïve Cohort: Placebo (N=31) | Flavivirus-naïve Cohort: PIZV 2 mcg (Low Dose) (N=31) | Flavivirus-naïve Cohort: PIZV 5 mcg (Medium Dose) (N=31) | Flavivirus-naïve Cohort: PIZV 10 mcg (High Dose) (N=32) | Flavivirus-primed Cohort: Placebo (N=36) | Flavivirus-primed Cohort: PIZV 2 mcg (Low Dose) (N=37) | Flavivirus-primed Cohort: PIZV 5 mcg (Medium Dose) (N=37) | Flavivirus-primed Cohort: PIZV 10 mcg (High Dose) (N=36)
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 1 | 1 | 1 | 3 | 2 | 2
Bronchitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 2 | 1 | 0 | 3 | 3 | 1
Dysuria (Renal and urinary disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2018-09-12): https://cdn.clinicaltrials.gov/large-docs/26/NCT03343626/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-26): https://cdn.clinicaltrials.gov/large-docs/26/NCT03343626/SAP_001.pdf